CLINICAL TRIAL: NCT05140668
Title: Comparison Between Supraclavicular And Infraclavicular Approach For Ultrasound-Guided Right Subclavian Venous Catheterization In Major Elective Surgeries And ICU Patients
Brief Title: Comparison Between Supraclavicular And Infraclavicular Approach For Right Subclavian Venous Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Maha Hamed Mohamed, Comparison between Supraclavicular And Infraclavicular Approach For Ultrasound-Guided Right Subclavian Venous Catheterization In Major Elective Surgeries And ICU Patients, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: soh-med-21-11-06
Record Dates: First submitted 2021-11-14; First posted 2021-12-01 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Central Line Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supraclavicular central venous catheterization approach group (Active Comparator): supraclavicular central venous catheterization group catheter is inserted in supraclavicular fossa (an indentation immediately above the clavicle) with a long-axis in plane approach
  Interventions: Device: Comparison between Supraclavicular And Infraclavicular Approach For Ultrasound-Guided Right Subclavian Venous Catheterization
- Infraclavicular central venous catheterization approach group (Active Comparator): infraclavicular central venous catheterization group catheter is inserted in infraclavicular fossa (an indentation, immediately below the clavicle, above the third rib and between the deltoid muscle laterally and medioclavicular line medially) with a short-axis out-of-plane approach
  Interventions: Device: Comparison between Supraclavicular And Infraclavicular Approach For Ultrasound-Guided Right Subclavian Venous Catheterization

INTERVENTIONS:
Device: Comparison between Supraclavicular And Infraclavicular Approach For Ultrasound-Guided Right Subclavian Venous Catheterization — Comparison between Supraclavicular And Infraclavicular Approach For Ultrasound-Guided Right Subclavian Venous Catheterization

SUMMARY:
A central venous catheter (CVC) is an indwelling device that is peripherally inserted into a larg central vein for a multitude of indications in major elective surgeries and ICU patients and now it's now with notable advance is the adjunct of ultrasound guidance, which has recently become the standard of care for CVCs placed in wanted site to decreases the complications

DETAILED DESCRIPTION:
A central venous catheter (CVC) is an indwelling device that is peripherally inserted into a large, central vein (most commonly the internal jugular, subclavian, or femoral) and advanced until the terminal lumen resides within the inferior vena cava, superior vena cava, or right atrium.for a multitude of indications including; total parenteral nutrition administration dialysis, plasmapheresis , medication administration, hemodynamic monitoring and to facilitate further complex interventions such as transvenous pacemaker placement inserted with Seldinger's technique. A notable advance is the adjunct of ultrasound guidance, which has recently become the standard of care for CVCs placed in wanted site owing to associated decreases in complications e.g. arterial puncture, haematoma formation, pneumothorax, haemothorax and catheterization failure and an increase in first-pass success.

ELIGIBILITY:
Inclusion criteria adult patients aged 20-79 y old who required central venous catheterization for : total parenteral nutrition administration dialysis plasmapheresis medication administration hemodynamic monitoring

Exclusion Criteria:

* Patient refusel Irritable patient Infection at the puncture site medical devices (chemoport, pacemaker,etc.) at the puncture site. right subclavian venous thrombosis haemostatic disorders current anticoagulant medication prescriptions previous history of surgery that might distort the anatomy of the right subclavian vein.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
to compare between the Supraclavicular and infraclavicular approach in right subclavian vein catheterization as regard accessibility sonar guided and number of punctures which is needed and the time of the procedure | 7 months
  After successful venous puncture, catheterization was attempted with the Seldinger's technique The guidewire and dilator were inserted to a depth of 10-15 cm and to the depth of venous puncture, respectively.
  We considered an attempt at catheterization as 'failed' if successful catheterization was not achieved within 3 min or If an anesthetist failed to catheterize the patient successfully within three attempts in 210 patients

SECONDARY OUTCOMES:
to compare complications which result from supraclavicular or approaches for right subclavian venous catheter insertion | 7 months
  monitoring of complications which can result from any of the two approaches e.g. arterial puncture, haematoma formation, pneumothorax, haemothorax it can monitored Clinically , blood gases and Chest X-Ray in 210 patients

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Beheshti MV. A concise history of central venous access. Tech Vasc Interv Radiol. 2011 Dec;14(4):184-5. doi: 10.1053/j.tvir.2011.05.002. PMID 22099008
- [Background] Konner K. History of vascular access for haemodialysis. Nephrol Dial Transplant. 2005 Dec;20(12):2629-35. doi: 10.1093/ndt/gfi168. Epub 2005 Oct 4. PMID 16204277
- [Background] American Society of Anesthesiologists Task Force on Central Venous Access; Rupp SM, Apfelbaum JL, Blitt C, Caplan RA, Connis RT, Domino KB, Fleisher LA, Grant S, Mark JB, Morray JP, Nickinovich DG, Tung A. Practice guidelines for central venous access: a report by the American Society of Anesthesiologists Task Force on Central Venous Access. Anesthesiology. 2012 Mar;116(3):539-73. doi: 10.1097/ALN.0b013e31823c9569. No abstract available. PMID 22307320
- [Background] Suess EM, Pinsky MR. Hemodynamic Monitoring for the Evaluation and Treatment of Shock: What Is the Current State of the Art? Semin Respir Crit Care Med. 2015 Dec;36(6):890-8. doi: 10.1055/s-0035-1564874. Epub 2015 Nov 23. PMID 26595049